CLINICAL TRIAL: NCT01845857
Title: A National Study of the Chronic Disease Self-Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kate Lorig, professor emertius, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SU-07212010-6585; 18933 IRB Protocol
Record Dates: First submitted 2010-08-09; First posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus, Type 2; Chronic Disease
Keywords: Long term health problems; chronic disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chronic Disease Self-Management Workshop (Experimental): Longitudinal study of participants who take the CDSMP workshop
  Interventions: Behavioral: Chronic Disease Self-Management Workshop

INTERVENTIONS:
Behavioral: Chronic Disease Self-Management Workshop — 6 week, small group self-management workshop

SUMMARY:
This survey will address important research, practice, and policy questions: How does Chronic Disease Self-Management Program (CDSMP) impact participants' general health, their health behaviors, and their need for health care utilization? Who benefits most from the CDSMP program? Are predicted gains maintained over a six and twelve month period? Can critical clinical changes be seen for those who are diabetic?

DETAILED DESCRIPTION:
A national survey of participant outcomes is important for documenting how the CDSMP program is impacting people with chronic diseases and influencing health care outcomes. This study will help bridge the research to practice gap and further our knowledge about the outcomes of evidence?based programs that are widely disseminated.

Investigators hope to learn the answers to the following questions for English and Spanish-speaking populations:

1. How does the CDSMP impact a person's general health?
2. Does the CDSMP increase the use of healthful behaviors?
3. Does the CDSMP impact health care utilization?
4. What are the characteristics of those who benefit from the CDSMP?
5. Can these benefits be maintained over 6 and 12 month periods?
6. For people with type 2 diabetes, and hemoglobin A1c be impacted by the CDSMP?

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Has a chronic health condition
* Attending a Chronic Disease Self-Management Workshop at a designated host site in the United states
* Speaks English or Spanish
* For blood test portion of study: have type 2 diabetes

Exclusion Criteria:

* Do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1170 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in Health Status (symptoms, activities limitations) | Baseline to 6 months
Change in Health Status (symptoms, activities limitations) | baseline to 12 months

SECONDARY OUTCOMES:
Change in Health behaviors (exercise, medical adherence) | baseline to 6 months
Change in health related quality of life | baseline to 6 months
Change in Metabolic control (HbA1c for type 2 diabetics) | baseline to 6 months
Change in Health Care Utilization | baseline to 6 months
  MD, emergency, hospital times and total nights
Change in Health behaviors (exercise, medical adherence) | baseline to 12 months
Change in health related quality of life | baseline to 12 months
Change in Metabolic control (HbA1c for type 2 diabetics) | baseline to 12 months
Change in Health Care Utilization | baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kate R Lorig, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Lorig KR, Ritter P, Stewart AL, Sobel DS, Brown BW Jr, Bandura A, Gonzalez VM, Laurent DD, Holman HR. Chronic disease self-management program: 2-year health status and health care utilization outcomes. Med Care. 2001 Nov;39(11):1217-23. doi: 10.1097/00005650-200111000-00008. PMID 11606875
- [Background] Lorig KR, Ritter PL, Gonzalez VM. Hispanic chronic disease self-management: a randomized community-based outcome trial. Nurs Res. 2003 Nov-Dec;52(6):361-9. doi: 10.1097/00006199-200311000-00003. PMID 14639082